CLINICAL TRIAL: NCT02594449
Title: A Pharmacodynamic and Safety Study of Benzalkonium Chloride Solution Clearing the Oral Colonized Bacterium in Healthy Volunteers
Brief Title: A Pharmacodynamic and Safety Study of BCS in Healthy Volunteers
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Lustre Pharmaceutical Lab Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: LC-PHB1505
Record Dates: First submitted 2015-10-29; First posted 2015-11-03 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-10

CONDITIONS: Healthy Volunteers
Keywords: Pharmacodynamic Study of BCS

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- low concentration Benzalkonium Chloride (Active Comparator): To use low concentration Benzalkonium Chloride Solution to gargle
  Interventions: Drug: Benzalkonium Chloride Solution
- high concentration Benzalkonium Chloride (Active Comparator): To use high concentration Benzalkonium Chloride Solution to gargle
  Interventions: Drug: Benzalkonium Chloride Solution
- Normal Saline (Placebo Comparator): To use Normal Saline to gargle
  Interventions: Drug: Benzalkonium Chloride Solution

INTERVENTIONS:
Drug: Benzalkonium Chloride Solution — To compare pharmacodynamics among the different concentrations of BCS and NS
  Other Names: Youkeshi

SUMMARY:
To compare pharmacodynamics among the different concentrations of BCS and NS.

DETAILED DESCRIPTION:
2 times mouthwash in the morning and at night. To collect bacterium samples to assess the pharmacodynamics among the different concentrations of BCS and NS: observe the changes of aerobic bacterial colonization in oropharyngeal over time during 24 hours, and assess the improvement of oral healthy status and the subjective feelings after 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers, males or females.
* Females with U-HCG negative.
* Signed ICFs, and could conduct this study with investigators.

Exclusion Criteria:

* History of mouthwash allergies, allergic rhinitis or dermatitis.
* Volunteers with oral ulcers, severe periodontal disease, oral mucosal lesions or oral cancer.
* Volunteers with removable denture.
* Had received special oral clean.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-10; Primary Completion 2016-01 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
The changes of aerobic bacterial colonization in oropharyngeal | 24 hours
  To collect the throat swab samples and supragingival plaque samples before and post administration, respectively, a total of 11 time points.

SECONDARY OUTCOMES:
The improvement of oral healthy status | 24 hours
  To use Plaque Index (PLI) to reflect volunteers' oral healthy status.
The volunteers' feelings | 24 hours
  The feelings including: comfortable, general comfortable, uncomfortable.

CONTACTS AND LOCATIONS:
Overall Officials: Shiyue Li, Professor, Principal Investigator — The First Affiliated Hospital of Guangzhou Medical University
Locations (1):
- The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China